CLINICAL TRIAL: NCT02788734
Title: Patient Reported Outcomes Measures (PROM) in Carpal Tunnel Therapies in Patients With Inherited Neuropathies
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Rochester (Other); University of Iowa (Other)
Responsible Party: Sponsor
Other Study IDs: INC6612; U01TR001263 (NIH)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2017-03

CONDITIONS: Carpal Tunnel Syndrome; Charcot-Marie-Tooth Disease; Inherited Peripheral Neuropathy
Keywords: carpal tunnel syndrome; CTS; inherited peripheral neuropathy; Charcot-Marie-Tooth disease; Hereditary Neuropathy; Pressure Palsies; CMT; HNPP
MeSH Terms: conditions — Carpal Tunnel Syndrome; Charcot-Marie-Tooth Disease; Inherited Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INC Contact Registry: INC Contact Registry will complete the online questionnaires
  Interventions: Other: Web-based survey

INTERVENTIONS:
Other: Web-based survey — This study protocol consists of one anonymous survey. Each participant can complete only one survey. The survey will take approximately 25 minutes to complete. The survey is designed to identify items that best reflect the symptom severity and functional status in patients with CTS and CMT. A unique link to the survey will be included in an email invitation distributed to all adult CMT or HNPP patients self-registered in the RDCRN INC Contact Registry. Upon clicking the link, the participant will be directed to the IRB-approved online consent form. Upon providing consent, the participant will be directed to the online survey.

SUMMARY:
The purpose of this study is to learn about focal compressive median neuropathy at the wrist (Carpal Tunnel Syndrome) and outcomes of therapies (e.g. conservative and surgery) in the upper extremities of patients diagnosed with an inherited neuropathy. All patients enrolled in the Rare Diseases Clinical Research Network (RDCRN) Inherited Neuropathies Consortium (INC) Contact Registry who have marked one of the following disorders: CMT1A, CMT1B, CMT2A, CMT4, CMTX, other known CMT peripheral neuropathy, other unknown CMT peripheral neuropathy, or Hereditary Neuropathy with liability to Pressure Palsies (HNPP), will be invited via email to participate in this online study.

DETAILED DESCRIPTION:
An online survey will be used to assess outcomes in conservative and surgical therapies used for carpal tunnel syndrome (CTS) in patients with a diagnosis of inherited neuropathy such as CMT or HNPP (Charcot-Marie-Tooth disease and Hereditary Neuropathy with liability to Pressure Palsies respectively). HNPP is an inherited neuropathy which is allelic to CMT1A. This patient reported outcome measurement will also assess symptom severity and functional status related to carpal tunnel syndrome (CTS) in various types of patients with inherited neuropathy.

The survey incorporates two validated questionnaires for the evaluation of outcomes related to carpal tunnel syndrome. The Boston Carpal Tunnel Questionnaire (BCTQ) is very specific to carpal tunnel syndrome (CTS). The Disability of Arm, Shoulder and Hand (DASH) questionnaire is less specific for CTS but has been shown to have equal validity in the assessment of outcomes in CTS. The relative non-specificity of DASH for CTS can be useful in assessing the possible contribution of CMT to the overall upper extremity symptom severity and functional outcome. Data collected from participants with a diagnosis or therapies for CTS can be compared to data collected from participants with no diagnosis or therapies for CTS.

Furthermore, the study will incorporate components from the CMTNS to assess the extent of CMT disease in the participants.

It is proposed that a retrospective analysis of patients with CMT who have symptoms in the upper extremities suggestive of carpal tunnel syndrome. Two validated questionnaires exploring changes in symptoms and functional status (BCTQ and DASH) can be used in evaluating outcomes of patients with reported symptoms or diagnosis of carpal tunnel syndrome.

The Boston Carpal Tunnel Questionnaire (BCTQ) is a 19 item scale which was developed specifically for carpal tunnel syndrome and consists of 11 questions to assess symptom severity and 8 questions to assess functional status. BCTQ has established test-retest reliability with a good Pearson's correlation of scores on re-test (0.91 for the symptoms severity component and 0.93 for the functional status component of the test). High internal consistency has also been reported for the BCTQ (0.88-9.92). Convergent validity has been demonstrated with high correlation between pre- and postoperative BCTQ scores and physical measures such as grip, key pinch and three-jaw pinch. Responsiveness of the BCTQ after carpal tunnel surgery has been demonstrated in randomized clinical trial settings. BCTQ has also been reported to be 2-4 times more responsive to clinical improvement in comparison to measures of neuromuscular impairment. High response rates have been reported with BCTQ with 80-93% at 6-12 weeks follow-up and between 67-93% at 6-12 months follow-up after carpal tunnel release. Response rates remained high at 85% at 2 years follow-up. Mailed follow-up response rate of 69% has been reported with a mean follow-up of 4.8 years. The mean time to complete BCTQ has been reported to be 5.6 minutes. There is no data to indicate the precision of BCTQ in relation to carpal tunnel syndrome.

The Disability of Arm, Shoulder and Hand (DASH) questionnaire is a 30 item scale which assesses symptoms and physical function. This questionnaire is not specific for carpal tunnel and can be used for a variety of disorders affecting the upper limb. DASH is intended to measure disability through an emphasis on upper extremity activity. The test-retest reliability of DASH has been demonstrated with a Pearson's 8 correlation of 0.9 in a group of patients with carpal tunnel syndrome.

The validity of DASH was demonstrated through correlation with BCTQ. Pre- and postoperative DASH scores also correlate with physical measures such as grip, key pinch and three-jaw pinch. Responsiveness through improved DASH scores has been demonstrated at three and six months post-surgery follow-up. BCTQ was found to be more responsive to DASH for carpal tunnel syndrome. Postal mail response rates have been shown to be 80-93% at 6-12 weeks and 66-98% at 6 months after carpal tunnel release. The mean time to complete DASH is reported to be 6.8 minutes. There is no data to indicate the precision of DASH in relation to carpal tunnel syndrome.

The survey data will be stored by the Rare Diseases Clinical Research Network's Data Management and Coordinating Center (DMCC) at the University of South Florida. Names or other personal health information will not be collected. Upon conclusion of the study period, the data will be sent to Dr. Michael Shy, principal investigator of the Inherited Neuropathies Consortium. Deidentified data will be sent to the database of Genotypes and Phenotypes (dbGaP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CMT or HNPP
* Adults age 18 years and older
* Self-Registration at the Inherited Neuropathies Consortium (INC) Contact Registry

Exclusion Criteria:

* Inability to provide informed consent and complete survey
* Inability to read or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The online survey will target adult CMT patients who have self-registered at the RDCRN Inherited Neuropathies Consortium (INC) Contact Registry, a web based contact registry developed and supported by the RDCRN Data Management and Coordinating Center (DMCC), located at the University of South Florida.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11-19 (Actual); Study Completion 2016-11-19 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | 2 months
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a 19 item scale which was developed specifically for carpal tunnel syndrome and consists of 11 questions to assess symptom severity and 8 questions to assess functional status
The Disability of Arm, Shoulder and Hand (DASH) questionnaire | 2 months
  30 item scale which assesses symptoms and physical function

CONTACTS AND LOCATIONS:
Overall Officials: David Herrmann, MBBCh, Study Chair — University of Rochester; Michael Shy, MD, Study Chair — University of Iowa; Callyn A Kirk, MSPH, Study Chair — USF Health Informatics Institute; Francis Panosyan, MD, PhD, Study Chair — University of Rochester
Locations (1):
- University of South Florida Health Informatics Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMillan CR, Binhammer PA. Which outcome measure is the best? Evaluating responsiveness of the Disabilities of the Arm, Shoulder, and Hand Questionnaire, the Michigan Hand Questionnaire and the Patient-Specific Functional Scale following hand and wrist surgery. Hand (N Y). 2009 Sep;4(3):311-8. doi: 10.1007/s11552-009-9167-x. Epub 2009 Mar 4. PMID 19259747
- [Background] Hobby JL, Venkatesh R, Motkur P. The effect of psychological disturbance on symptoms, self-reported disability and surgical outcome in carpal tunnel syndrome. J Bone Joint Surg Br. 2005 Feb;87(2):196-200. doi: 10.1302/0301-620x.87b2.15055. PMID 15736742
- [Background] Harder K, Lukschu S, Dunda SE, Krapohl BD. Results after simple decompression of the ulnar nerve in cubital tunnel syndrome. GMS Interdiscip Plast Reconstr Surg DGPW. 2015 Dec 21;4:Doc19. doi: 10.3205/iprs000078. eCollection 2015. PMID 26734540
- [Background] Katz JN, Fossel KK, Simmons BP, Swartz RA, Fossel AH, Koris MJ. Symptoms, functional status, and neuromuscular impairment following carpal tunnel release. J Hand Surg Am. 1995 Jul;20(4):549-55. doi: 10.1016/S0363-5023(05)80265-5. PMID 7594277
- [Background] Kaye JJ, Reynolds JM. Carpal tunnel syndrome: using self-report measures of disease to predict treatment response. Am J Orthop (Belle Mead NJ). 2007 Apr;36(4):E59-62. PMID 17703268
- [Background] Wintman BI, Winters SC, Gelberman RH, Katz JN. Carpal tunnel release. Correlations with preoperative symptomatology. Clin Orthop Relat Res. 1996 May;(326):135-45. PMID 8620634
- [Background] Murphy SM, Herrmann DN, McDermott MP, Scherer SS, Shy ME, Reilly MM, Pareyson D. Reliability of the CMT neuropathy score (second version) in Charcot-Marie-Tooth disease. J Peripher Nerv Syst. 2011 Sep;16(3):191-8. doi: 10.1111/j.1529-8027.2011.00350.x. PMID 22003934
- [Background] Greenslade JR, Mehta RL, Belward P, Warwick DJ. Dash and Boston questionnaire assessment of carpal tunnel syndrome outcome: what is the responsiveness of an outcome questionnaire? J Hand Surg Br. 2004 Apr;29(2):159-64. doi: 10.1016/j.jhsb.2003.10.010. PMID 15010164
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Earle N, Zochodne DW. Is carpal tunnel decompression warranted for HNPP? J Peripher Nerv Syst. 2013 Dec;18(4):331-5. doi: 10.1111/jns5.12047. PMID 24171697
- [Background] Stahl S, Blumenfeld Z, Yarnitsky D. Carpal tunnel syndrome in pregnancy: indications for early surgery. J Neurol Sci. 1996 Mar;136(1-2):182-4. doi: 10.1016/0022-510x(95)00335-y. PMID 8815170
- [Background] Arthur-Farraj PJ, Murphy SM, Laura M, Lunn MP, Manji H, Blake J, Ramdharry G, Fox Z, Reilly MM. Hand weakness in Charcot-Marie-Tooth disease 1X. Neuromuscul Disord. 2012 Jul;22(7):622-6. doi: 10.1016/j.nmd.2012.02.008. Epub 2012 Mar 28. PMID 22464564
- [Background] Potocki L, Chen KS, Koeuth T, Killian J, Iannaccone ST, Shapira SK, Kashork CD, Spikes AS, Shaffer LG, Lupski JR. DNA rearrangements on both homologues of chromosome 17 in a mildly delayed individual with a family history of autosomal dominant carpal tunnel syndrome. Am J Hum Genet. 1999 Feb;64(2):471-8. doi: 10.1086/302240. PMID 9973284
- [Background] Pareyson D, Marchesi C. Diagnosis, natural history, and management of Charcot-Marie-Tooth disease. Lancet Neurol. 2009 Jul;8(7):654-67. doi: 10.1016/S1474-4422(09)70110-3. PMID 19539237
- [Background] Harding AE, Thomas PK. The clinical features of hereditary motor and sensory neuropathy types I and II. Brain. 1980 Jun;103(2):259-80. doi: 10.1093/brain/103.2.259. PMID 7397478
- [Background] Miller MJ, Williams LL, Slack SL, Nappi JF. The hand in Charcot-Marie-Tooth disease. J Hand Surg Br. 1991 May;16(2):191-6. doi: 10.1016/0266-7681(91)90175-n. PMID 2061663
- [Background] Azmaipairashvili Z, Riddle EC, Scavina M, Kumar SJ. Correction of cavovarus foot deformity in Charcot-Marie-Tooth disease. J Pediatr Orthop. 2005 May-Jun;25(3):360-5. doi: 10.1097/01.bpo.0000150807.90052.98. PMID 15832156
- [Background] Sraj SA, Saghieh S, Abdulmassih S, Abdelnoor J. Medium to long-term follow-up following correction of pes cavus deformity. J Foot Ankle Surg. 2008 Nov-Dec;47(6):527-32. doi: 10.1053/j.jfas.2008.06.007. PMID 19239862
- [Background] Faldini C, Traina F, Nanni M, Mazzotti A, Calamelli C, Fabbri D, Pungetti C, Giannini S. Surgical treatment of cavus foot in Charcot-Marie-tooth disease: a review of twenty-four cases: AAOS exhibit selection. J Bone Joint Surg Am. 2015 Mar 18;97(6):e30. doi: 10.2106/JBJS.N.00794. PMID 25788311
- [Background] Dreher T, Hagmann S, Wenz W. Reconstruction of multiplanar deformity of the hindfoot and midfoot with internal fixation techniques. Foot Ankle Clin. 2009 Sep;14(3):489-531. doi: 10.1016/j.fcl.2009.06.001. PMID 19712887
- [Result] Kotsis SV, Chung KC. Responsiveness of the Michigan Hand Outcomes Questionnaire and the Disabilities of the Arm, Shoulder and Hand questionnaire in carpal tunnel surgery. J Hand Surg Am. 2005 Jan;30(1):81-6. doi: 10.1016/j.jhsa.2004.10.006. PMID 15680560
- [Result] Gay RE, Amadio PC, Johnson JC. Comparative responsiveness of the disabilities of the arm, shoulder, and hand, the carpal tunnel questionnaire, and the SF-36 to clinical change after carpal tunnel release. J Hand Surg Am. 2003 Mar;28(2):250-4. doi: 10.1053/jhsu.2003.50043. PMID 12671856
- [Result] Kadzielski J, Malhotra LR, Zurakowski D, Lee SG, Jupiter JB, Ring D. Evaluation of preoperative expectations and patient satisfaction after carpal tunnel release. J Hand Surg Am. 2008 Dec;33(10):1783-8. doi: 10.1016/j.jhsa.2008.06.019. PMID 19084178
- [Result] Beaton DE, Katz JN, Fossel AH, Wright JG, Tarasuk V, Bombardier C. Measuring the whole or the parts? Validity, reliability, and responsiveness of the Disabilities of the Arm, Shoulder and Hand outcome measure in different regions of the upper extremity. J Hand Ther. 2001 Apr-Jun;14(2):128-46. PMID 11382253
- [Result] Niekel MC, Lindenhovius AL, Watson JB, Vranceanu AM, Ring D. Correlation of DASH and QuickDASH with measures of psychological distress. J Hand Surg Am. 2009 Oct;34(8):1499-505. doi: 10.1016/j.jhsa.2009.05.016. Epub 2009 Aug 22. PMID 19703733
- [Result] Ebersole GC, Davidge K, Damiano M, Mackinnon SE. Validity and responsiveness of the DASH questionnaire as an outcome measure following ulnar nerve transposition for cubital tunnel syndrome. Plast Reconstr Surg. 2013 Jul;132(1):81e-90e. doi: 10.1097/PRS.0b013e318290faf6. PMID 23806957
- [Result] Jarvik JG, Comstock BA, Heagerty PJ, Haynor DR, Fulton-Kehoe D, Kliot M, Franklin GM. Magnetic resonance imaging compared with electrodiagnostic studies in patients with suspected carpal tunnel syndrome: predicting symptoms, function, and surgical benefit at 1 year. J Neurosurg. 2008 Mar;108(3):541-50. doi: 10.3171/JNS/2008/108/3/0541. PMID 18312102
- [Result] Eklund E, Svensson E, Hager-Ross C. Hand function and disability of the arm, shoulder and hand in Charcot-Marie-Tooth disease. Disabil Rehabil. 2009;31(23):1955-62. doi: 10.1080/09638280902874170. PMID 19479509
- [Result] Appleby MA, Neville-Smith M, Parrott MW. Functional outcomes post carpal tunnel release: a modified replication of a previous study. J Hand Ther. 2009 Jul-Sep;22(3):240-8; quiz 249. doi: 10.1016/j.jht.2009.03.001. Epub 2009 May 19. PMID 19457636
- [Result] Jarvik JG, Comstock BA, Kliot M, Turner JA, Chan L, Heagerty PJ, Hollingworth W, Kerrigan CL, Deyo RA. Surgery versus non-surgical therapy for carpal tunnel syndrome: a randomised parallel-group trial. Lancet. 2009 Sep 26;374(9695):1074-81. doi: 10.1016/S0140-6736(09)61517-8. PMID 19782873
- [Result] Verdugo RJ, Salinas RA, Castillo JL, Cea JG. Surgical versus non-surgical treatment for carpal tunnel syndrome. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD001552. doi: 10.1002/14651858.CD001552.pub2. PMID 18843618
- [Result] Atroshi I, Hofer M, Larsson GU, Ornstein E, Johnsson R, Ranstam J. Open compared with 2-portal endoscopic carpal tunnel release: a 5-year follow-up of a randomized controlled trial. J Hand Surg Am. 2009 Feb;34(2):266-72. doi: 10.1016/j.jhsa.2008.10.026. PMID 19181226
- [Result] Maggard MA, Harness NG, Chang WT, Parikh JA, Asch SM, Nuckols TK; Carpal Tunnel Quality Group. Indications for performing carpal tunnel surgery: clinical quality measures. Plast Reconstr Surg. 2010 Jul;126(1):169-179. doi: 10.1097/PRS.0b013e3181da8685. PMID 20595866
- [Result] Adkinson JM, Zhong L, Aliu O, Chung KC. Surgical Treatment of Cubital Tunnel Syndrome: Trends and the Influence of Patient and Surgeon Characteristics. J Hand Surg Am. 2015 Sep;40(9):1824-31. doi: 10.1016/j.jhsa.2015.05.009. Epub 2015 Jun 30. PMID 26142079
- [Result] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Result] Videler AJ, Beelen A, van Schaik IN, de Visser M, Nollet F. Limited upper limb functioning has impact on restrictions in participation and autonomy of patients with hereditary motor and sensory neuropathy 1a. J Rehabil Med. 2009 Sep;41(9):746-50. doi: 10.2340/16501977-0419. PMID 19774309
- [Result] Videler AJ, Beelen A, Aufdemkampe G, de Groot IJ, Van Leemputte M. Hand strength and fatigue in patients with hereditary motor and sensory neuropathy (types I and II). Arch Phys Med Rehabil. 2002 Sep;83(9):1274-8. doi: 10.1053/apmr.2002.34282. PMID 12235608